CLINICAL TRIAL: NCT04703803
Title: Treatment of Myofascial Pain Syndrome With Lidocaine Injection in Patients With Cancer in Palliative Care: a Randomized Clinical Trial
Brief Title: Efficacy of Myofascial Pain Syndrome Treatment in Patients With Cancer in Palliative Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nereida Kilza da Costa Lima, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPS_palliativecancer
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Myofascial Pain Syndromes; Cancer
Keywords: Myofascial Pain Syndromes; Cancer Pain; Palliative care
MeSH Terms: conditions — Myofascial Pain Syndromes; Neoplasms; Cancer Pain | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Randomized, comparative, single-blinded interventional study
Who Masked: Outcomes Assessor
Masking Description: A member of the research team who doesn´t know whether the participant is in the intervention or control group will be responsible for the reassessment (after 72 hours and 1 week) to measure the outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% lidocaine injection (Experimental): The intervention group will be submitted to the trigger point injection procedure with 1% lidocaine (the sum of all needled trigger points will have a maximum of 10 ml), in a single intervention
  Interventions: Combination Product: 1% lidocaine injection in trigger points
- Control Group (No Intervention): The control group will receive usual care, defined as the treatment for pain prescribed by their assistant doctors.

INTERVENTIONS:
Combination Product: 1% lidocaine injection in trigger points — The trigger point injection procedure with 1% lidocaine will be e (the sum of all needled trigger points will have a maximum of 10 ml), in a single intervention
  Arms: 1% lidocaine injection

SUMMARY:
Palliative Care is active holistic care offered to people who are in intense suffering related to their health, resulting from a serious life-threatening illness, with a focus on improving the quality of life. Among the symptoms that cause suffering, physical pain has a prominent role in terms of prevalence and impact on well-being, especially in the subgroup of patients with terminal cancer. Myofascial Pain Syndrome may be one of the components of pain in cancer patients in palliative care. However, the literature is scarce in defining the prevalence of this condition in this population, and there is no evidence of the benefit of needling treatment with 1% lidocaine in these patients until now. The objectives of this study are to determinate the prevalence of myofascial pain syndrome and to evaluate the effectiveness of myofascial pain treatment with 1% lidocaine injection in reducing pain in palliative cancer patients, comparing it with a control group in usual care.

DETAILED DESCRIPTION:
This is a clinical trial designed as a comparative, randomized, single-blinded intervention study. Patients will be recruited from wards and radiotherapy sector of the Ribeirão Preto Clinical Hospital - Ribeirão Preto Medical School, University of São Paulo (FMRP-USP). Initially, patients aged 50 years or older with cancer in palliative care will be evaluated to assess the prevalence of myofascial pain syndrome using Travel and Simons' diagnostic criteria and for the following variables: demographic characteristics, functional status (Palliative Performance Scale), pain intensity (visual analog scale and pain threshold measurement with a pressure gauge), prognostic score (Palliative Prognosis Score), depression and anxiety (Hospital Anxiety and Depression Scale), quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 PAL) and analgesic drugs in use. The participants that (1) accomplish the Travel and Simons' diagnostic criteria for myofascial pain syndrome, (2) have performance status on the Karnofsky scale of 30 or more, and (3) have pain intensity on visual analog scale of 5 or more will be randomized for the clinical trial. The sample size calculation resulted in 15 participants for each group, totaling a sample composed of 30 patients. The intervention group will be submitted to the trigger point injection procedure with 1% lidocaine, and the control group will receive usual care, defined as the treatment for pain prescribed by their assistant doctors. Both groups will be reevaluated after 72 hours and 1 week after the procedure. In the analysis statistics, chi-square test (or Fisher's exact test) will be used to evaluate categorical variables. For the comparison between the groups at each moment (before and after intervention) will be used the linear mixed effects model. The significance level established was <0.05. SAS Statistical Software (version 9.3; SAS Institute, Inc. Cary , NC) will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants that

  1. accomplish the Travel and Simons' diagnostic criteria for myofascial pain syndrome,
  2. have pain intensity on visual analog scale of 5 or more,
  3. have performance status on the Karnofsky Performance Status scale of 30 or more.

Exclusion Criteria:

* Use of high dose anticoagulants (RNI above the therapeutic range);
* Patients with hemorrhagic diathesis;
* Patients with moderate to severe dementia syndrome;
* Patients with diagnosis of acute confusional state during the follow-up;
* Occurrence of clinical complication or intervention that could compromise the reevaluation of pain in the following days (for example, undergoing a surgical procedure or nerve block) or death.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | 72 hours and 7 days
  Assessed by Visual Analogic Scale (0 to 10). This evaluation will be collected at baseline, after 72 hours and after 7 days in follow-up.

SECONDARY OUTCOMES:
Change in pain threshold measurement | 72 hours and 7 days
  Assessed with a pressure gauge (Kg). This evaluation will be collected at baseline, after 72 hours and after 7 days in follow-up.
Change in number of analgesic drugs in use | 72 hours and 7 days
  Evaluation of the number of drugs in use, if there was an increase, reduction or maintenance of the number and doses of analgesic drugs comparing to the baseline.
Assessment of depression and anxiety simptoms | 7 days
  Assessed by Hospital Anxiety and Depression Scale- scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. Higher scores mean worse outcome.
Assessment of quality of life | 7 days
  Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnarie Core 15 PAL

CONTACTS AND LOCATIONS:
Locations (1):
- Laís Araujo Dos Santos Vilar, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD to be made available after the end of the study protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of results of study
Access Criteria: Researchers after the review and approval of protocol by the principal investigator

REFERENCES:
- [Derived] Santos-Vilar LAD, Freitas-Passos IF, Rossi BM, Blauth FG, Pontes VCB, Moriguti JC, Riberto M, Lima NKDC. Lidocaine Needling in Myofascial Pain Syndrome for Palliative Oncologic Care: A Randomized Clinical Study. J Palliat Med. 2024 Jul;27(7):888-894. doi: 10.1089/jpm.2023.0641. Epub 2024 Mar 14. PMID 38484328
- See also: Webpage of the Ribeirão Preto Medical School — http://fmrp.usp.br